CLINICAL TRIAL: NCT00811603
Title: Optimal Timing for Antibiotic Prophylaxis for Elective Cesarean Delivery in Term Gestations: A Randomized, Controlled Trial Comparing Cefazolin Administration Prior to Skin Incision Versus Following Cord Clamping
Brief Title: Trial Comparing the Optimal Timing of Antibiotic Prophylaxis at the Time of Cesarean Delivery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MemorialCare (Other)
Collaborators: University of California, Irvine (Other)
Responsible Party: Leo Pevzner, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 474-07
Record Dates: First submitted 2008-12-17; First posted 2008-12-19 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Cesarean Section; Infection
Keywords: Antibiotic; Prophylaxis; Cesarean; Infection; Antibiotic prophylaxis
MeSH Terms: conditions — Infections | interventions — Cefazolin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Patients who receive antibiotic prophylaxis after clamping of the umbilical cord
  Interventions: Drug: Cefazolin (Timing of Antibiotic Prophylaxis)
- 2 (Experimental): Patients who receive antibiotic prophylaxis prior to skin incision
  Interventions: Drug: Cefazolin (Timing of Antibiotic Prophylaxis)

INTERVENTIONS:
Drug: Cefazolin (Timing of Antibiotic Prophylaxis) — Patients scheduled for a cesarean delivery will be randomly assigned to receive Cefazolin (antibiotic prophylaxis) either prior to skin incision or after the clamping of the umbilical cord

SUMMARY:
The purpose of this study is to evaluate the rates of maternal and neonatal infectious morbidity in gravid patients undergoing cesarean delivery. Specifically, the investigators are examining whether the timing of antibiotic administration has any effect on rates of maternal and neonatal infections, neonatal sepsis work-up and length of hospital stay.

DETAILED DESCRIPTION:
Nearly fifty years have passed since Burke et al first demonstrated in animal model the reduction of infection rates in contaminated skin incisions with administration of antibiotic prophylaxis. Further research in the area confirmed the benefit of prophylactic antibiotics in human subjects. Patients who develop surgical infections are 60% more likely to spend time in intensive care unit, five times more likely to be readmitted to the hospital, and have twice the mortality rate compared to patients without infections. As a result the potential health care costs are staggering. Recently, the National Surgical Infection Prevention Project endorsed the recommendation that antibiotic prophylaxis should be administered within 60 minutes before skin incision. This model has been universally accepted in all surgical fields with the exception of obstetrics.

Cesarean delivery has been shown to be the most important risk factor for post-partum maternal infection. In fact, women undergoing cesarean delivery have a five to twenty-fold greater risk for developing infection compared to those undergoing vaginal delivery. Recent review by Cochrane Database found that there is an inconsistent and variable application of current recommendations in regard to appropriate timing, administration and choice of drug used for antibiotic prophylaxis at the time of cesarean delivery. Cesarean section holds a unique position amongst all the surgical procedures as being the only one where prophylactic antibiotics are administered after the incision is made. The concern for intrapartum fetal exposure of prophylactic antibiotics suppressing microbial growth and thereby masking neonatal sepsis led to a tradition of delaying antibiotic administration until umbilical cord clamping. While a recent study demonstrated that antibiotic levels do indeed reach therapeutic levels within cord blood very quickly after administration to the mother, no adverse outcomes to the newborns have ever been documented as a result. To date only four studies have looked at the timing of prophylactic administration at the time of cesarean section.

In 1982, Cunningham et al randomized 642 women "at high risk for infection following cesarean delivery" to receiving antibiotics before or after cord clamping. The authors demonstrated that there was no difference between uterine infection rates between the two groups. While significantly more infants exposed to intrapartum maternal antibiotics were evaluated for sepsis, there were no cases of neonatal bacteremia in either group. However, it should be noted that the pediatricians in this study were fully aware of whether antibiotics had been given before or after cord clamping. Wax et al revisited the issue by randomizing 90 consecutive term women in labor to receiving cefazolin preoperatively or after skin incision. While the authors failed to show any statistical significance between two groups, this study was clearly underpowered as only four cases achieved primary outcomes. Furthermore, the authors failed to demonstrate a significant increase is suspected sepsis in newborns whose mothers received cefazolin preoperatively. In 2005, Thigpen et al once again demonstrated that there was no disadvantage to the infant in regard to infectious morbidity. In addition, there was no difference in maternal infectious morbidity regardless of when antibiotics were administered. However, the results are questionable as nearly a quarter of all subjects received penicillin for GBS prophylaxis. Finally, Sullivan included 357 women in a well designed randomized, double-blinded study that demonstrated a statistically significant reduction in maternal infectious morbidity when the antibiotics where administered preoperatively. Not only was there no difference between two groups in regard to neonatal infection, but there was actually significantly fewer NICU admission days in preoperative antibiotic group.

Despite the evidence that preoperative prophylactic antibiotics pose no harm to the fetus, obstetrics has been slow to adopt this practice. It is no wonder that cesarean infection rates have been shown to be considerably higher than comparable surgical procedures. While the evidence clearly demonstrates the absence of negative impact of preoperative antibiotics on neonatal outcomes, a contemporary scientific evaluation of the reduction in maternal infectious morbidity is warranted before adopting this practice on universal basis.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Any patient at term (>37 weeks gestation) undergoing a scheduled cesarean delivery

Exclusion Criteria:

* Women younger than 18 years
* Patients who are febrile during or prior to screening or with a diagnosis of clinical suspicion of endometritis (with or without maternal fever)
* Patients who present with ruptured membranes
* Known fetal malformations
* Contraindications to cefazolin administration (known anaphylactic reaction to penicillins or known cephalosporin allergy)
* Any exposure to antibiotics in one week prior to cesarean delivery
* Obstetrical indication for an emergent cesarean delivery
* Patients taking glucocorticoids or other immunosuppressant therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-08; Primary Completion 2009-06 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To assess the rates of maternal infectious morbidity with preoperative administration of antibiotics when compared to antibiotic prophylaxis given following umbilical cord clamping | 6 weeks

SECONDARY OUTCOMES:
To assess incidence of neonatal infectious morbidity (i.e. rates of sepsis work-up, confirmed sepsis, and length of hospital stay) between two study arms | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Chan, MD, Principal Investigator — Memorial Medical Center
Locations (2):
- United States (2):
  - Long Beach Memorial Medical Center, Long Beach, California
  - University of California, Irvine Medical Center, Orange, California